CLINICAL TRIAL: NCT04398550
Title: Specific Carbohydrate Diet vs. Mediterranean Diet Therapy in Ulcerative Colitis - A Clinical Trial
Brief Title: SCD vs. Mediterranean Diet Therapy in Ulcerative Colitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hamed Khalili, Assistant Professor of Medicine at Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P000298
Record Dates: First submitted 2020-02-24; First posted 2020-05-21 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis
Keywords: Diet
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The investigators, subjects, and remaining study staff will not be intentionally unblinded. Due to the nature of the study, subjects, study staff, and investigators interacting with the subjects will likely be able to figure out what diet the subject is assigned to, however, the exact diet will not be explicitly revealed to them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific Carbohydrate Diet (Experimental): Exclusive consumption of the specific carbohydrate diet for 6 weeks
  Interventions: Other: Specific Carbohydrate Diet
- Mediterranean Diet (Experimental): Exclusive consumption of the Mediterranean diet for 6 weeks
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Specific Carbohydrate Diet — Diet restricts all but simple carbohydrates and allows for inclusion of fresh fruits, vegetables, unprocessed meats, and homemade lactose-free cheese and yogurt.
  Arms: Specific Carbohydrate Diet
Other: Mediterranean Diet — Diet rich in whole vegetables, fruit, plant-based protein, and olive oil, with moderate amounts of seafood and dairy, and limited in sugar-sweetened goods, red meat, and nutrients like heme and sodium.
  Arms: Mediterranean Diet

SUMMARY:
Although patients and physicians have shown tremendous interest in the effect of diet on ulcerative colitis, there is a lack of significant evidence for providers to make practical recommendations with. In this study, the investigators hope to find out if dietary therapy by either the Specific Carbohydrate Diet (SCD) or the Mediterranean diet will help improve ulcerative colitis symptoms for patients with mild to moderately active disease. In addition, the investigators will compare disease activity and changes in the intestinal bacterial composition in the colon that occur with the Mediterranean or the SCD diet in active ulcerative colitis.

This study is proposed as a single-site randomized trial consisting of 10 study visits to Massachusetts General Hospital (MGH) over 12 weeks. Participants in this study will be randomly assigned to the SCD or Mediterranean diet. The investigators ask that participants exclusively consume their assigned diet for 6 weeks, with all meals and snacks prepared by the metabolic kitchen within MGH. Participants will need to pick up food from MGH every 5-7 days, and will meet with a study dietitian before they begin and weekly during the diet therapy.

There will be a screening visit to determine eligibility for the study, as well as study visits at weeks 0, 1, 2, 4, 6, and a 10 week follow-up at MGH, in which participants will fill out questionnaires. Participants will need to provide stool samples at screening, week 6, and week 10. In addition, blood will be drawn at week 0 and week 6, and if participants are getting a clinically-indicated colonoscopy at the time of screening, up to eight research biopsies may be collected during the procedure.

DETAILED DESCRIPTION:
This randomized, parallel-group feeding study will examine the influence of Mediterranean and SCD diets on gut microbiota, luminal inflammation, and disease-specific clinical indices in patients with mild to moderate ulcerative colitis (UC). 50 patients will be randomized to follow either the SCD or Mediterranean diet in a 1:1 ratio. Once informed consent is obtained, subjects will enter a 2-week screening period. Eligible subjects will be enrolled in the feeding treatment for 6 weeks followed by an additional follow-up visit at 10 weeks (4 weeks after feeding treatment completion). The total time to complete the study is 12 weeks. The metabolic kitchen within the Metabolism and Nutrition Research Center at MGH Translational and Clinical Research (TCRC) Unit will be responsible for preparing and packaging food for participants to pick up, as well as performing all necessary nutritional assessments. Participants will be provided with 3 meals and 2 snacks a day during the 6-week dietary intervention. Patient menus will be identical in each diet and will rotate on a 3-day basis. Total calories for each diet will be tailored according to each participant's body composition.

ELIGIBILITY:
Inclusion Criteria:

* History of active ulcerative colitis for at least 3 months before screening
* Ulcerative colitis confirmed by colonoscopy or flexible sigmoidoscopy within 2 years of screening
* Mild to moderate ulcerative colitis at the time of screening (2 < Mayo score < 12)
* 1 ≤ Endoscopy subscore ≤ 2, or fecal calprotectin > 150 mcg/g within 2 weeks of screening
* Patients on 5-aminosalicylates (e.g. mesalamine, etc.) must be on a stable dose for ≥ 4 weeks prior to screening
* Patients on treatment with immunosuppressive (azathioprine/6-mercaptopurine and methotrexate) or biologic medications (infliximab, adalimumab, and golimumab) must be on stable dose for 8 weeks prior to baseline
* At the time of baseline, patients may be on no more than 20 mg of prednisone and 9 mg of budesonide MMX

Exclusion Criteria:

* Patients with Crohn's disease or indeterminate colitis
* History of colectomy
* Presence of ileal pouch or ostomy
* History of colonic dysplasia
* Evidence of active bacterial or viral gastroenteritis as indicated by positive stool studies for ova & parasites, clostridium difficile, and stool culture
* Severe to fulminant colitis
* Recent hospitalizations (within 2 weeks of screening) for ulcerative colitis requiring IV steroids
* Recent systemic antibiotics use (within 2 weeks of screening)
* Presence of the following labs indicative of severe colitis: a. Hemoglobin < 8.0 g/dl b. Albumin < 3.0 g/dl
* Use of Total Parenteral Nutrition (TPN)
* Active use of anti-diarrheal medications
* Use of cyclosporine, tacrolimus, or thalidomide within 2 months prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Partial Mayo Clinic Score | Week 6
  The partial Mayo clinic score measures disease activity, on a scale of 0 to 9. The higher scores indicate more severe disease activity (the worse outcome).

SECONDARY OUTCOMES:
Partial Mayo Clinic Score | Week 1, Week 2, Week 4, Week 10 follow-up
  The partial Mayo clinic score measures disease activity, on a scale of 0 to 9. The higher scores indicate more severe disease activity (the worse outcome).
Inflammatory Bowel Disease Questionnaire (IBDQ10) | Week 1, Week 2, Week 4, Week 6, and Week 10 follow-up
  The IBDQ10 measures quality of life, on a scale of 10 to 70. The higher scores indicate a better outcome (better quality of life).
Short Form (12) Health Survey (SF-12) | Week 1, Week 2, Week 4, Week 6, and Week 10 follow-up
  The SF-12 measures health-related quality of life, split into physical and mental health scores on a scale of 0 to 100. The higher scores indicate a better outcome.
Simple Clinical Colitis Activity Index (SCCAI) | Week 1, Week 2, Week 4, Week 6, and Week 10 follow-up
  The SCCAI measures disease activity, on a scale of 0 to 21. The higher scores indicate a worse outcome (more severe disease activity).
stool microbiome | Week 6 and Week 10 follow-up
  Stool samples will be taken at screening/baseline and week 6 and 10 to assess change in fecal microbiome pattern, measured using R2Aspread plating, QiagenAllPrep RNA/DNA Mini kit, and whole genome shotgun sequencing.
fecal calprotectin | Week 6 and Week 10 follow-up
  Stool samples will be taken at screening/baseline and week 6 and 10 to assess change in fecal calprotectin levels.
C-reactive protein | Week 6
  Blood will be drawn at baseline and week 6 to assess change in C-reactive protein levels.

CONTACTS AND LOCATIONS:
Overall Officials: Hamed Khalili, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified information may be shared with other collaborators and entities involved in generating data.

REFERENCES:
- [Background] Albenberg LG, Wu GD. Diet and the intestinal microbiome: associations, functions, and implications for health and disease. Gastroenterology. 2014 May;146(6):1564-72. doi: 10.1053/j.gastro.2014.01.058. Epub 2014 Feb 4. PMID 24503132
- [Background] Ferguson A, Sedgwick DM, Drummond J. Morbidity of juvenile onset inflammatory bowel disease: effects on education and employment in early adult life. Gut. 1994 May;35(5):665-8. doi: 10.1136/gut.35.5.665. PMID 8200562
- [Background] Poullis A, Foster R, Shetty A, Fagerhol MK, Mendall MA. Bowel inflammation as measured by fecal calprotectin: a link between lifestyle factors and colorectal cancer risk. Cancer Epidemiol Biomarkers Prev. 2004 Feb;13(2):279-84. doi: 10.1158/1055-9965.epi-03-0160. PMID 14973103
- [Background] Martinez-Medina M, Denizot J, Dreux N, Robin F, Billard E, Bonnet R, Darfeuille-Michaud A, Barnich N. Western diet induces dysbiosis with increased E coli in CEABAC10 mice, alters host barrier function favouring AIEC colonisation. Gut. 2014 Jan;63(1):116-24. doi: 10.1136/gutjnl-2012-304119. Epub 2013 Apr 18. PMID 23598352
- [Background] Stenman LK, Holma R, Eggert A, Korpela R. A novel mechanism for gut barrier dysfunction by dietary fat: epithelial disruption by hydrophobic bile acids. Am J Physiol Gastrointest Liver Physiol. 2013 Feb 1;304(3):G227-34. doi: 10.1152/ajpgi.00267.2012. Epub 2012 Nov 29. PMID 23203158
- [Background] Lee D, Albenberg L, Compher C, Baldassano R, Piccoli D, Lewis JD, Wu GD. Diet in the pathogenesis and treatment of inflammatory bowel diseases. Gastroenterology. 2015 May;148(6):1087-106. doi: 10.1053/j.gastro.2015.01.007. Epub 2015 Jan 15. PMID 25597840
- [Background] Jowett SL, Seal CJ, Pearce MS, Phillips E, Gregory W, Barton JR, Welfare MR. Influence of dietary factors on the clinical course of ulcerative colitis: a prospective cohort study. Gut. 2004 Oct;53(10):1479-84. doi: 10.1136/gut.2003.024828. PMID 15361498
- [Background] Magee EA, Edmond LM, Tasker SM, Kong SC, Curno R, Cummings JH. Associations between diet and disease activity in ulcerative colitis patients using a novel method of data analysis. Nutr J. 2005 Feb 10;4:7. doi: 10.1186/1475-2891-4-7. PMID 15705205
- [Background] Degagne E, Pandurangan A, Bandhuvula P, Kumar A, Eltanawy A, Zhang M, Yoshinaga Y, Nefedov M, de Jong PJ, Fong LG, Young SG, Bittman R, Ahmedi Y, Saba JD. Sphingosine-1-phosphate lyase downregulation promotes colon carcinogenesis through STAT3-activated microRNAs. J Clin Invest. 2014 Dec;124(12):5368-84. doi: 10.1172/JCI74188. Epub 2014 Oct 27. PMID 25347472
- [Background] Jantchou P, Morois S, Clavel-Chapelon F, Boutron-Ruault MC, Carbonnel F. Animal protein intake and risk of inflammatory bowel disease: The E3N prospective study. Am J Gastroenterol. 2010 Oct;105(10):2195-201. doi: 10.1038/ajg.2010.192. Epub 2010 May 11. PMID 20461067
- [Background] Liang J, Nagahashi M, Kim EY, Harikumar KB, Yamada A, Huang WC, Hait NC, Allegood JC, Price MM, Avni D, Takabe K, Kordula T, Milstien S, Spiegel S. Sphingosine-1-phosphate links persistent STAT3 activation, chronic intestinal inflammation, and development of colitis-associated cancer. Cancer Cell. 2013 Jan 14;23(1):107-20. doi: 10.1016/j.ccr.2012.11.013. Epub 2012 Dec 27. PMID 23273921
- [Background] Ijssennagger N, Belzer C, Hooiveld GJ, Dekker J, van Mil SW, Muller M, Kleerebezem M, van der Meer R. Gut microbiota facilitates dietary heme-induced epithelial hyperproliferation by opening the mucus barrier in colon. Proc Natl Acad Sci U S A. 2015 Aug 11;112(32):10038-43. doi: 10.1073/pnas.1507645112. Epub 2015 Jul 27. PMID 26216954
- [Background] IJssennagger N, Derrien M, van Doorn GM, Rijnierse A, van den Bogert B, Muller M, Dekker J, Kleerebezem M, van der Meer R. Dietary heme alters microbiota and mucosa of mouse colon without functional changes in host-microbe cross-talk. PLoS One. 2012;7(12):e49868. doi: 10.1371/journal.pone.0049868. Epub 2012 Dec 11. PMID 23239972
- [Background] Zimmermann MB, Chassard C, Rohner F, N'goran EK, Nindjin C, Dostal A, Utzinger J, Ghattas H, Lacroix C, Hurrell RF. The effects of iron fortification on the gut microbiota in African children: a randomized controlled trial in Cote d'Ivoire. Am J Clin Nutr. 2010 Dec;92(6):1406-15. doi: 10.3945/ajcn.110.004564. Epub 2010 Oct 20. PMID 20962160
- [Background] Werner T, Wagner SJ, Martinez I, Walter J, Chang JS, Clavel T, Kisling S, Schuemann K, Haller D. Depletion of luminal iron alters the gut microbiota and prevents Crohn's disease-like ileitis. Gut. 2011 Mar;60(3):325-33. doi: 10.1136/gut.2010.216929. Epub 2010 Nov 12. PMID 21076126
- [Background] Kleinewietfeld M, Manzel A, Titze J, Kvakan H, Yosef N, Linker RA, Muller DN, Hafler DA. Sodium chloride drives autoimmune disease by the induction of pathogenic TH17 cells. Nature. 2013 Apr 25;496(7446):518-22. doi: 10.1038/nature11868. Epub 2013 Mar 6. PMID 23467095
- [Background] Wu C, Yosef N, Thalhamer T, Zhu C, Xiao S, Kishi Y, Regev A, Kuchroo VK. Induction of pathogenic TH17 cells by inducible salt-sensing kinase SGK1. Nature. 2013 Apr 25;496(7446):513-7. doi: 10.1038/nature11984. Epub 2013 Mar 6. PMID 23467085
- [Background] Yosef N, Shalek AK, Gaublomme JT, Jin H, Lee Y, Awasthi A, Wu C, Karwacz K, Xiao S, Jorgolli M, Gennert D, Satija R, Shakya A, Lu DY, Trombetta JJ, Pillai MR, Ratcliffe PJ, Coleman ML, Bix M, Tantin D, Park H, Kuchroo VK, Regev A. Dynamic regulatory network controlling TH17 cell differentiation. Nature. 2013 Apr 25;496(7446):461-8. doi: 10.1038/nature11981. Epub 2013 Mar 6. PMID 23467089
- [Background] HAAS SV, HAAS MP. The treatment of celiac disease with the specific carbohydrate diet; report on 191 additional cases. Am J Gastroenterol. 1955 Apr;23(4):344-60. No abstract available. PMID 14361377
- [Background] Halmos EP, Christophersen CT, Bird AR, Shepherd SJ, Gibson PR, Muir JG. Diets that differ in their FODMAP content alter the colonic luminal microenvironment. Gut. 2015 Jan;64(1):93-100. doi: 10.1136/gutjnl-2014-307264. Epub 2014 Jul 12. PMID 25016597
- [Background] Lindsay JO, Whelan K, Stagg AJ, Gobin P, Al-Hassi HO, Rayment N, Kamm MA, Knight SC, Forbes A. Clinical, microbiological, and immunological effects of fructo-oligosaccharide in patients with Crohn's disease. Gut. 2006 Mar;55(3):348-55. doi: 10.1136/gut.2005.074971. Epub 2005 Sep 14. PMID 16162680
- [Background] Halmos EP, Christophersen CT, Bird AR, Shepherd SJ, Muir JG, Gibson PR. Consistent Prebiotic Effect on Gut Microbiota With Altered FODMAP Intake in Patients with Crohn's Disease: A Randomised, Controlled Cross-Over Trial of Well-Defined Diets. Clin Transl Gastroenterol. 2016 Apr 14;7(4):e164. doi: 10.1038/ctg.2016.22. PMID 27077959
- [Background] De Filippo C, Cavalieri D, Di Paola M, Ramazzotti M, Poullet JB, Massart S, Collini S, Pieraccini G, Lionetti P. Impact of diet in shaping gut microbiota revealed by a comparative study in children from Europe and rural Africa. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14691-6. doi: 10.1073/pnas.1005963107. Epub 2010 Aug 2. PMID 20679230
- [Background] Obih C, Wahbeh G, Lee D, Braly K, Giefer M, Shaffer ML, Nielson H, Suskind DL. Specific carbohydrate diet for pediatric inflammatory bowel disease in clinical practice within an academic IBD center. Nutrition. 2016 Apr;32(4):418-25. doi: 10.1016/j.nut.2015.08.025. Epub 2015 Nov 30. PMID 26655069
- [Background] Suskind DL, Cohen SA, Brittnacher MJ, Wahbeh G, Lee D, Shaffer ML, Braly K, Hayden HS, Klein J, Gold B, Giefer M, Stallworth A, Miller SI. Clinical and Fecal Microbial Changes With Diet Therapy in Active Inflammatory Bowel Disease. J Clin Gastroenterol. 2018 Feb;52(2):155-163. doi: 10.1097/MCG.0000000000000772. PMID 28030510